CLINICAL TRIAL: NCT02987764
Title: Neurodevelopmental Outcomes of Cord Milking in Preterm Infants: Randomized Controlled Trial
Brief Title: Cord Milking Impacts Neurodevelopmental Outcomes in Very Low Birth Weight Infants
Acronym: Cordmilking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Subject recruitment and enrollment was low throughout the three years the study was active.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Meena Garg, MD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 15-001134
Record Dates: First submitted 2016-12-01; First posted 2016-12-09 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Very Low Birth Weight Infant
Keywords: Premature; Birth weight
MeSH Terms: conditions — Premature Birth; Birth Weight | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cord Milking (Experimental): The research team member will untwist the cord, and hold it in a vertical position. The cord will then be milked twice towards the abdominal insertion of the cord. The cord will be cut 1 inch above the abdominal wall. After milking for exact measurement of the cord will be obtained.
  Interventions: Other: cord milking
- Observational (No Intervention): Observational infants will receive usual care with immediate cord clamping by the delivering obstetrician. The time of cord clamping will be recorded for both groups using a timer.

INTERVENTIONS:
Other: cord milking — For infants in the cord milking group, the cord will be clamped at the longest distance possible and neonatal team will bring the infant to the resuscitation table for further care. The clinical care will be provided by the clinicians taking care of the infant. The research team will be trained and be responsible for requesting the obstetrician in advance to provide the maximum length of umbilical cord.
  Arms: Cord Milking

SUMMARY:
Premature birth is a major risk factor for perinatal brain damage and cerebral palsy (CP) with 47% of all CP cases occurring in infants with birth weight less than 2500 g. CP has life-long neurological consequences that affect quality of life for the patient. In the last 2 decades, improvements in neonatal intensive care have improved survival of VLBW infants significantly. This increased survival of VLBW infants poses new challenges towards developing novel treatments and interventions to decrease neurodevelopmental impairment and CP. While it is common for extremely preterm infant to survive at 23 weeks of gestation, the neurologic consequences range from learning difficulties and cognitive defects to severe disability and cerebral palsy. Currently prenatal neuroprotective agents such as corticosteroids are utilized whenever a preterm birth is anticipated. However, there are no proven postnatal interventions to prevent brain damage and cerebral palsy in VLBW infants.

Many recent studies show that delaying umbilical cord clamping (DCC) may improve hemodynamic stability and decrease intraventricular hemorrhage (IVH) in preterm infants. A decrease in incidence of IVH has a conceivable prospective benefit of decreasing brain injury and improving long-term outcomes. Based on these findings, the American College of Obstetricians and Gynecologist and American Academy of Pediatrics endorse that DCC may benefit the preterm infants. However, these recommendations have not been adopted by most obstetricians in USA. The main concern regarding the practice of DCC is the care delay in initiating resuscitation and providing the needed care to this vulnerable population.

Therefore, as an alternative to DCC, method of cord milking (CM) has been developed to provide cord blood transfusion to premature infants. CM offers a more practical alternative to delayed cord clamping that may provide the same benefits without the need to delay resuscitation. However, there are very few studies of CM in VLBW infants and there is no evidence demonstrating long-term neurological outcomes and CP after CM.

The investigators hypothesize that cord milking in VLBW infants will result in improving cerebral oxygenation, function and result in improved long-term neurodevelopmental outcomes at 2 years of post-menstrual age. Premature infants born at less than or equal to 32 weeks gestation age will receive cord milking after cutting versus standard care of immediate cord clamping.

DETAILED DESCRIPTION:
Primary Aims

To Measure:

1. Cerebral oxygenation and function (aEEG abnormalities) in first 24 hours of life
2. Neurodevelopmental outcomes at 18 - 24 months PMA Secondary Aims

1. Assessment of Improved transition: Delivery room resuscitation, Apgar scores, acidosis from cord gas or first hour blood gas 2. Neurological injury assessment: IVH/PVIH/PVL on head ultrasound on day #3-5 and day #7-14, and at 36 wk PMA, MRI at 36 wk CGA 3. CVS response: Blood pressure and ionotropic support in first 3-5 days 4. Hematological assessment: Hemoglobin, Hematocrit of admission, and first 72 hours of life, need for phototherapy and highest bilirubin level in first 7 days, blood transfusions needed till 36 wk PMA 5. Gastrointestinal protection: Necrotizing enterocolitis till 36 wk PMA In this pilot study, we plan to enroll 15 VLBW infants in each group (n=30) from Mattel Children's Hospital and Santa Monica Hospital labor and delivery. Data pertaining to primary and secondary aims will be obtained from EMR. Follow up utilizing Bayley's scores of infant development (BSID III) will be scheduled at 18-22 months PMA

ELIGIBILITY:
Inclusion Criteria:

* 1. Expected delivery at <32 week GA.

Exclusion Criteria:

* 1. Prenatal diagnosis of chromosomal or severe congenital malformations such as cyanotic congenital heart disease 2. Cord accidents such as ruptured Vasa Previa results in fetal blood loss, need for urgent delivery, placental abruption and cord prolapse 3. considered non-viable by attending neonatologist or obstetrician 4. Consent not granted

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2016-05; Primary Completion 2018-05-15 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Measure Cerebral oxygenation and function | First 24 hours of life

SECONDARY OUTCOMES:
Apgar Scores | 1 and 5 minutes
  Basic score to measure the newborn status. From 0 to 10.
Neurological injury assessment | Days 3-5 and at 36 weeks postmenstrual age
  Head ultrasound on day #3-5
Neurological injury assessment | weeks postmenstrual age
  MRI at 36 wk CGA
Hematological assessment | First 72 hours of life
  Hematocrit of admission
Gastrointestinal protection | 36 weeks postmenstrual age
  Necrotizing enterocolitis till 36 wk PMA
Measure Neurodevelopmental impairment | 18-24 months postmenstrual age
  Outcome assessments will be conducted by physicians or nurse practitioners or occupation therapist specializing in neonatal follow-up examination using Bayley Scales of Infant Development III

CONTACTS AND LOCATIONS:
Locations (1):
- Mattel Children's Hospital UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No